CLINICAL TRIAL: NCT06366711
Title: Remote Antenatal Maternal-fetal Telemedicine Monitoring in High-risk Pregnancies: a Feasibility and Acceptability Study
Brief Title: Remote Telemedicine Fetal Monitoring Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Collaborators: GE Healthcare (Industry); Nestmedic Spolka Akcyjna (Industry)
Responsible Party: Principal Investigator, Jack Hamer, Clinical research fellow in maternal-fetal medicine, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23/BW/MAT/NO/754
Record Dates: First submitted 2024-03-28; First posted 2024-04-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy, High Risk; Telemonitoring; Telemedicine; Ultrasound; Cardiotocography

STUDY DESIGN:
Intervention Model Description: 15 participants split in to three arms. The sample size has been determined as a pragmatic sample taking into consideration the needs of the feasibility study to meet the stated objectives as well as being achievable within the time and cost constraints of the study. 15 participants will ensure a thorough assessment of the stated objectives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Home antenatal CTG monitoring (Experimental): Participants will be asked to use the remote monitoring devices twice a week, on mutually agreed days for a minimum of 30 minutes each time. Ideally participants will use the home CTG monitor for at least a four-week period or until delivery.
  Interventions: Device: Pregnabit Pro device and PregnaOne platform
- Home antenatal ultrasound monitoring (Experimental): Participants will be asked to use the remote monitoring devices once a fortnight, on mutually agreed days for the duration by which the scan has been completed. Ideally participants will use the home ultrasound monitor for at least a 8-week period or until delivery.
  Interventions: Drug: Pulsenmore device
- Usage of both home antenatal ultrasound and CTG monitoring devices (Experimental): Follow both device plans above.
  Interventions: Device: Pregnabit Pro device and PregnaOne platform; Drug: Pulsenmore device

INTERVENTIONS:
Device: Pregnabit Pro device and PregnaOne platform — Remote CTG device for pregnancy care
  Arms: Home antenatal CTG monitoring; Usage of both home antenatal ultrasound and CTG monitoring devices
Drug: Pulsenmore device — Remote ultrasound device for pregnancy care
  Arms: Home antenatal ultrasound monitoring; Usage of both home antenatal ultrasound and CTG monitoring devices

SUMMARY:
During pregnancy, certain conditions may arise that mean regular monitoring of both mother and baby are needed to ensure timely interventions and avoid the need for further treatments. These situations include problems with high blood pressure, obstetric cholestasis (characterised by liver-related itchiness), preterm premature rupture of membranes (PPROM), and a history of stillbirth. Monitoring typically involves assessing the mother's blood pressure and urine, recording the baby's heart rate over a specific duration, and conducting regular ultrasound scans. Such monitoring can require frequent hospital visits, often multiple times a week, which can be very time consuming. More recently, new technology has emerged, enabling remote monitoring of mother and baby outside of the hospital setting, such as their own home. However, research on these technologies is still very limited.

Our study aims to address this research gap by inviting women with the above conditions to volunteer for home-based monitoring, alongside their routine hospital care. Participants will be divided into three groups: one group will use transducers, attached to the mothers tummy, to capture the baby's heartbeat; another group will use a handheld ultrasound device connected to their mobile phones, allowing them to observe the baby; and a third group will use both devices. All device information will be transmitted securely to the healthcare professional for analysis. The investigators aim to assess the feasibility of conducting remote monitoring of mother and baby, whilst understanding how acceptable the technology is received.

Importantly, the data collected will only be evaluated by the research team and will not be intended to influence patient's current planned antenatal care. Women will receive comprehensive training on the devices. The study will additionally gather feedback from participating women through questionnaires, both at the study's outset and its conclusion, regarding their experiences and emotions related to the research.

DETAILED DESCRIPTION:
The primary aim of this research proposal is to explore the feasibility and acceptability of home antenatal maternal-fetal monitoring technology within a high-risk pregnancy group. The investigators hypothesise that home monitoring is feasible and acceptable to pregnant women.

Pregnant women from 32+0 weeks' gestation onwards receiving regular outpatient antenatal care including routine ultrasound and CTG monitoring on the Day Assessment Unit (DAU) at the Birmingham Women's hospital (BWH). They will continue their regular antenatal care whilst using the devices.

* Home antenatal CTG monitoring using the Pregnabit Pro device and PregnaOne platform only - 5 participants.
* Home antenatal ultrasound monitoring using the Pulsenmore device only - 5 participants.
* Usage of both home antenatal ultrasound and CTG monitoring devices - 5 participants.

Following consent, participants will be provided with the home monitoring equipment including a face-to-face education session on their usage. A schedule for home monitoring will be agreed. Participants will be asked to complete a short questionnaire about their views and expectations of home telemetry, including some basic patient characteristics.

• Home CTG monitoring - Pregnabit Pro device and PregnaOne platform: Participants will be asked to use the remote monitoring devices twice a week, on mutually agreed days for a minimum of 30 minutes each time. Ideally participants will use the home CTG device for at least a four-week period or until delivery.

• Home ultrasound monitoring - Pulsenmore: Participants will be asked to use the remote monitoring devices fortnightly, on mutually agreed days . Ideally participants will use the home ultrasound device for at least a eight-week period or until delivery.

• Both home CTG and ultrasound monitoring: Participants will follow both above device plans as noted above

The recordings will be uploaded automatically and wirelessly to the respective online clinical dashboards, whereby two members of the research team will securely review the images contemporaneously.

End of participation:

Upon completion, equipment will be collected, and participants will be asked to complete a short exit questionnaire about the usability, reassurance, feelings of control and overall feedback. Additionally, patients will repeat the GAD-7 anxiety questionnaire.

End of study:

All data will be formally collated and analysed with respect to the above study outcomes, enabling the research team to retrieve an overall determination as to whether these devices are feasible and acceptable for the pregnancy population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years
* Gestational age 32+0 weeks onwards.
* Singleton pregnancy.
* Receiving antenatal care which includes routine antenatal fetal monitoring for one of the 4 index conditions (pregnancy induced hypertension (PIH), obstetric cholestasis, PPROM and previous history of stillbirth)
* Able to give written informed consent.
* Willing to attend hospital immediately in the event of an unexpected finding whilst using the home devices.

Exclusion Criteria:

* Multiple pregnancy.
* Fetal abnormalities or a non-viable fetus.
* Body mass index (BMI) ≥35
* Women with internal cardiac devices such as pacemaker and implantable cardioverter defibrillator.
* History of allergic reaction to skin adhesives and/or latex.
* Acute or chronic skin lesions and wounds in areas in contact with the device.
* Medical or midwifery concerns regarding maternal and/or fetal conditions such that inpatient care is recommended.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
The number of participants that produce interpretable fetal ultrasound scans for each episode of intermittent home monitoring. | Through study completion, an average of 6 months
  Ultrasound scans will be assessed upon the criterion that the device is currently licensed for: fetal movements, fetal heartbeat and an objective assessment of the liquor volume.
The number of participants that produce interpretable antenatal maternal-fetal monitoring cardiotocogram (CTG) traces for each episode of intermittent home monitoring. | Through study completion, an average of 6 months
  Completion of an at least 20 minutes of uninterrupted interpretable fetal heart recording which has computerised capability.

SECONDARY OUTCOMES:
The number of participants completing the full schedule of home maternal-fetal monitoring episodes. | Through study completion, an average of 6 months
  Number of monitoring episodes out of total episodes desired at study onset.
To explore how acceptability and participant views can best be assessed within a future clinical trial using wearable technology at home? | 6 months
  Questionnaires
The number of women approached who agreed to participate within the study. | Pre-intervention
  Number participants agreeing out of total women approached
What are the views of participants and healthcare professionals regarding acceptability of home maternal-fetal monitoring. | Pre-intervention
  Pre-intervention questionnaire using a 5 point Likert Scale (range from Strongly agree on the left, to strongly disagree on the right). No total score, each question individual and a tick box.
What are the views of participants and healthcare professional regarding acceptability of home maternal-fetal monitoring. | Immediately after the intervention
  Post-intervention questionnaire using a 5 point Likert Scale (range from Strongly agree on the left, to strongly disagree on the right). No total score, each question individual and a tick box.
What are the emotions of participants prior to and following usage of home maternal-fetal monitoring. | Pre-intervention
  Pre-intervention questionnaire using the accredited GAD-7 anxiety questionnaire. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
What are the emotions of participants prior to and following usage of home maternal-fetal monitoring. | Immediately after the intervention
  Post-intervention questionnaire using the accredited GAD-7 anxiety questionnaire. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
The number of participants with unexpected clinical outcomes detected whilst using home monitoring devices, which warrants patients to attend maternity triage for assessment and/or modification of ones antenatal care. | Through study completion, an average of 6 months
  Number of unexpected outcomes out of total number of monitoring episodes

CONTACTS AND LOCATIONS:
Overall Officials: Leo Gurney, Study Director — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham Women's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Vance J, Emms A, Hodgetts Morton V, Morris RK, Gurney L. Remote maternal-fetal telemedicine monitoring for high-risk pregnancy care: A feasibility study. PLoS One. 2025 Nov 14;20(11):e0336797. doi: 10.1371/journal.pone.0336797. eCollection 2025. PMID 41237146